CLINICAL TRIAL: NCT04731857
Title: Diagnostic Value of Exome and Genome Sequencing As Well As Conventional Methods in Rare Diseases and Familial Tumor Syndromes
Brief Title: Diagnostic Value of Exome/ Genome Sequencing, Conventional Methods in Rare Diseases and Familial Tumor Syndromes
Acronym: EXGEFATU
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: EXGEFATU
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rare Diseases; Genetic Predisposition
Keywords: Rare Diseases; Genetic Predisposition; Next Generation Sequencing (NGS); Polygenic risk scores (PRSs); Repeat-Expansion; Genetic variation
MeSH Terms: conditions — Rare Diseases; Genetic Predisposition to Disease; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Genetic diseases: For the retrospective data analysis, patients with genetic diseases of any age and, if available, other family members, for whom genetic analyzes were carried out between 10/2016 and 12/2020, should be included. This equates to approximately 13,000 records, minus combined analyzes in the same patient, an estimated 12,000 individuals.
  Interventions: Genetic: Retrospective data analysis

INTERVENTIONS:
Genetic: Retrospective data analysis — The outlined evaluation contributes to the improvement of molecular genetic diagnostics in patient care - for example when which diagnostics can be sensibly recommended for patients with which indications or not. Diagnostic gaps can be systematically evaluated and specifically addressed in the future. This potentially affects every examination assignment for current and future patients. In addition, the evaluation of the PRSs for example, can contribute significantly to the timely introduction to routine diagnostics. For familial breast cancer, according to the guidelines, there may be very specific preventive measures. Estimates currently assume up to 5% of patients, which would mean up to 25 cases per year with a potentially adapted management for patients with the question of a tumor disease alone.

SUMMARY:
For the retrospective data analysis, patients with genetic diseases of any age and, if available, other family members, for whom genetic analyzes were carried out between 10/2016 and 12/2020, should be included. This equates to approximately 13,000 records, minus combined analyzes in the same patient, an estimated 12,000 individuals.

DETAILED DESCRIPTION:
The methodological developments of the last few years allow the broad use of next-generation-sequencing (NGS) -based methods in the routine molecular genetic diagnosis of genetic diseases.The aim of the retrospective data analysis is to create a solid data basis for further discussion regarding the development and mapping of diagnostic algorithms and subsequent supply routes. For the genome data, this evaluation is to be expanded to include the evaluation of the Polygenic risk scores (PRSs) in the sense of an additional finding.

ELIGIBILITY:
Inclusion Criteria:

* Patient with genetic disease or
* Family members
* Genetic analysis between 10/2016 and 12/2020 at the Institute for Medical Genetics and Applied Genomics at the University Hospital Tübingen

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetic diseases of any age and, if present, other family members, for whom genetic analyzes were carried out between 10/2016 and 12/2020 at the Institute for Medical Genetics and Applied Genomics at the University Hospital Tübingen.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | Day 1
  Number of established probable diagnosis using molecular genetic diagnostics

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haack, Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No